CLINICAL TRIAL: NCT05799508
Title: Consequences of COVID-19 Infection for Child Health and Wellbeing: Protocol for a Prospective, Observational, Longitudinal Study in Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: ID 3777
Record Dates: First submitted 2023-03-29; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-02

CONDITIONS: Long COVID
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective follow-up of children with SARS-CoV-2

ELIGIBILITY:
Inclusion Criteria:

* Children aged 0-18 years
* The child sought/needed primary or secondary medical care for COVID-19
* Laboratory (RT-PCR,) [18]
* 28 days - 3 months from the onset of COVID-19 symptoms
* Parent's/carer's/guardian's consent to participate

Exclusion Criteria:

* adults

Ages: 4 Weeks to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population will consist of patients diagnosed with COVID-19 and admitted to the hospitals and/or assessed in primary care among our Institution. Patients will be identified from existing local cohorts.
  Inclusion criteria:
  * Children aged 0-18 years
  * The child sought/needed primary or secondary medical care for COVID-19
  * Laboratory (RT-PCR,) [18]
  * 28 days - 3 months from the onset of COVID-19 symptoms
  * Parent's/carer's/guardian's consent to participate The survey for paediatric follow-up is based on the previously developed adult questionnaire. The survey has been adapted to specific age groups to identify specific symptoms in children.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
number of children developing long covid | up to 36 months
  prevalence of post covid condition at 3-6-12-18-24-36 months after SARS-CoV-3 infection

SECONDARY OUTCOMES:
duration and characteristics of children with long covid, also according to variants | up to 36 months
  prevalence of post covid condition according to the original SARS-CoV-2 variant at 3-6-12-18-24-36 months after SARS-CoV-3 infection

CONTACTS AND LOCATIONS:
Locations (1):
- Gemelli, Roma, Italy

IPD SHARING:
Plan to Share IPD: Yes
to contact the PI, sharing planned with GBD
Supporting Information: Study Protocol, SAP, CSR